CLINICAL TRIAL: NCT03854942
Title: Opioid Modulation of the Effect of Alcohol on the Dopaminergic Reward System: a [18F]-Fallypride- and [18F]-Fluoro-DOPA-PET Study.
Brief Title: Study of the Opioid Modulation of the Effect of Alcohol on the Dopaminergic Reward System
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment rate could not be met in the study period, review group was dissolved before regular end of study. Recruitment was therefore terminated.
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 10-002
Record Dates: First submitted 2019-02-18; First posted 2019-02-26 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Addiction
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Arm (Other): 7 days placebo intake - i.v. injection of physiological saline solution (0,9%) - PET followed by 7 days placebo intake - i.v. injection of ethanol solution (6 Vol.-%) - PET
  Interventions: Drug: Placebo
- Second Arm (Other): 7 days placebo intake - i.v. injection of physiological saline solution (0,9%) - PET - 7 days naltrexone intake (Nemexin, 50 mg once daily during the first 2 days, 100 mg daily for the following 5 days) - injection of physiological saline solution (0,9%) - PET
  Interventions: Drug: Placebo; Drug: Naltrexone
- Third Arm (Other): 7 days placebo intake - i.v. injection of ethanol solution (6 Vol.-%) - PET - 7 days naltrexone (Nemexin, 50 mg once daily during the first 2 days, 100 mg daily for the following 5 days) intake - i.v. injection of ethanol solution (6 Vol.-%) - PET
  Interventions: Drug: Placebo; Drug: Naltrexone

INTERVENTIONS:
Drug: Placebo — Placebo oral tablet daily
Drug: Naltrexone — Naltrexone (Nemexin) oral tablet 50 mg daily for 2 days, Naltrexone (Nemexin) oral tablet 100 mg daily for 5 days
  Arms: Second Arm; Third Arm

SUMMARY:
About 10% of the calculable loss of health and quality of life in industrial countries can be attributed to excessive alcohol consumption. Behavioural pharmacological, genetic and clinical studies on alcohol dependence suggest a multifactorial model for the development of the disease, which ascribes an important role in the development of the disease to genetic variance, educational style and continued substance use. Animal and human experimental studies suggest that continued alcohol consumption leads to a pathological activation of the mesolimbic reward system. In the presented study, the modification of the alcohol-mediated activation of the mesolimbic reward system by the administration of the opiate antagonist naltrexone will be investigated in a human in vivo model. The aim is to gain important insights for the further development of pharmacological treatment options for alcohol dependence. Further development of pharmacological treatment options for alcohol dependence seems urgently necessary in order to slow down the high tendency to relapse and prolong the short abstinence period.

ELIGIBILITY:
Inclusion Criteria:

* age: 21-45 years
* The subject is able to understand the nature, extent and individual consequences of the clinical trial
* Maintained ability to give consent, certified by a psychiatrist (specialist)
* A personally dated informed consent form signed by the test participant
* No current and/or historical psychiatric disorder (secured by standardized psychiatric interview (DIAX: Composite International Diagnostic Interview))
* Non-smokers (no nicotine addiction within the last 6 months prior to sequential allocation)
* OPRM1 Asp40 carrier (functional polymorphism in amino acid residue 40 of μ-opioid receptor gene (OPRM1)) (in AC for inclusion in first and third treatment arm)
* Highly effective contraception method with a failure rate of <1%: Hormonal contraceptive methods (oral: "contraceptive pill", incl. combined oral contraceptives; subcutaneous implants; injectable contraceptives); intrauterine pessary, vasectomy of the partner, tube ligation ("sterilisation") or sexual abstinence
* Persons who are legally competent and mentally able to understand and follow the instructions of the study staff
* MRI capability

Exclusion Criteria:

* hypersensitivity to the investigational product or a chemically similar substance or component of the investigational product
* Participation in other clinical trials during or within 6 months prior to this clinical trial
* Medical or psychological circumstances which may jeopardise the proper conduct of the clinical trial
* Physical illnesses which could interfere with the planned examinations according to their type and severity, could have an influence on the parameters to be examined or could endanger the volunteer during the course of the examination
* Inability to adhere to the study protocol
* Limited or completely revoked legal capacity
* Acute suicidal tendency or external hazard
* Poor overall condition
* Participation in a study using ionising radiation in the last five years.
* Regular medication (e.g. MAO inhibitors)
* Alcohol abuse, alcohol dependency or addiction illness / abuse of addictive substances in history
* Existence of other exclusion criteria for participation in MRI examinations (non-removable metal parts in the body, left-handedness, pacemakers)
* Known hypersensitivity to carbidopa or any of the other components
* Relevant organic diseases: in particular: Narrow angle glaucoma, vascular diseases, central nervous neurological diseases; body weight of more than 150 kg (contraindications PET - scan)
* Clinically significant deviations in clinical chemistry or haematology or clinically significant abnormalities
* Melanoma-specific skin lesions or anamnesis of a previous melanoma disease
* Persons who are accommodated in an establishment by court order or official order
* Persons who are dependent on or have an employment relationship with the sponsor or investigator

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Pharmacological effect of naltrexone on the dopamine synthesis rate of a healthy OPRM1 Asp40-bearing men under the influence of alcohol measured with [18F]-fluoro-DOPA PET. | 28 days
Dopamine D2 receptor availability in the structures of the ventral and dorsal striatum of a healthy µ-opioid receptor gen (OPRM1, Asp40 Allel)-bearing men under the influence of alcohol measured with [18F]-fallypride Positron Emission Tomography. | 28 days

SECONDARY OUTCOMES:
Pharmacological effect of ethanol on dopamine D2 receptor availability in healthy men measured with [18F]-fallypride Positron Emission Tomography. | 28 days
Pharmacological effect of ethanol on the dopamine synthesis rate of the ventral and dorsal striatum in healthy men measured with [18F]-fluoro-DOPA PET. | 28 days
Pharmacological effect of Naltrexone on dopamine D2 receptor availability in healthy men measured with [18F]-fallypride Positron Emission Tomography. | 28 days
Pharmacological effect of Naltrexone on the dopamine synthesis rate of ventral and dorsal striatum in healthy men measured with [18F]-fluoro-DOPA PET. | 28 days

OTHER OUTCOMES:
Modulation of extrastriatal dopamine D2/D3 receptor availability measured with [18F]-fallypride in structures of the anterior cingulum using Positron Emission Tomography. | 28 days
Relationship between impulsive behaviour and functionality of the dopamine synthesis rate and dopamine D2 receptor availability | 28 days
  Evaluation of impulsive behaviour using BIS (Barratt Impulsiveness Scale) questionnaire
Relationship between impulsive behaviour and functionality of the dopamine synthesis rate and dopamine D2 receptor availability | 28 days
  Evaluation of impulsive behaviour using Neo-FFI (NEO-Fünf-Faktoren-Inventar) questionnaire
Relationship between impulsive behaviour and functionality of the dopamine synthesis rate and dopamine D2 receptor availability | 28 days
  Evaluation of impulsive behaviour using I7 (Impulsivitätsfragebogen (impulsivity questionnaire) nach Eysenck) questionnaire
Interaction between subjective alcohol effects and placebo/naltrexone effects | 28 days
  Exploratively, the interaction between subjective alcohol effects and placebo/naltrexone effects will be investigated using VAS (visual analogue scale of alcoholic desire) questionnaire.
Interaction between subjective alcohol effects and placebo/naltrexone effects | 28 days
  Exploratively, the interaction between subjective alcohol effects and placebo/naltrexone effects will be investigated using OCDS (Obsessive Compulsive Drinking Scale) questionnaire.
Interaction between subjective alcohol effects and placebo/naltrexone effects | 28 days
  Exploratively, the interaction between subjective alcohol effects and placebo/naltrexone effects will be investigated using ESA (Erfassung subjektiver Alkoholwirkungen (Determination of subjective alcohol effects)) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No